CLINICAL TRIAL: NCT03405935
Title: A Phase 3b, Multicenter, Open-Label Study to Evaluate Switching From an Elvitegravir/Cobicistat/Emtricitabine/Tenofovir Alafenamide Fixed-Dose Combination Regimen or a Tenofovir Disoproxil Fumarate Containing Regimen to Fixed-Dose Combination of Bictegravir/Emtricitabine/Tenofovir Alafenamide in Elderly, Virologically-Suppressed, HIV-1 Infected Subjects Aged ≥ 65 Years
Brief Title: Study to Evaluate Switching From an E/C/F/TAF Fixed-Dose Combination (FDC) Regimen or a TDF Containing Regimen to B/F/TAF FDC in Human Immunodeficiency Virus-1 (HIV-1) Infected Participants Aged ≥ 65 Years
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-380-4449; 2017-003428-61 (EudraCT Number)
Record Dates: First submitted 2018-01-12; First posted 2018-01-23 (Actual); Results first posted 2019-12-05 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-11

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- B/F/TAF (Experimental): B/F/TAF FDC for at least 96 weeks.
  Interventions: Drug: B/F/TAF

INTERVENTIONS:
Drug: B/F/TAF — 50/200/25 mg FDC tablet administered orally once daily without regard to food.
  Other Names: Biktarvy®

SUMMARY:
The primary objective of this study is to characterize the virologic efficacy of switching virologically suppressed participants on an elvitegravir/cobicistat/emtricitabine/tenofovir alafenamide (E/C/F/TAF) fixed-dose combination (FDC) regimen or a tenofovir disoproxil fumarate (TDF) containing regimen to bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF) FDC.

ELIGIBILITY:
Key Inclusion Criteria:

* Currently receiving an antiretroviral regimen of E/C/F/TAF FDC (or emtricitabine [FTC]/TDF + 3rd agent if currently or previously participated in Study GS-US-292-1826 [NCT02616783]) for ≥ 3 months
* Documented plasma HIV-1 ribonucleic acid (RNA) < 50 copies/mL during treatment with E/C/F/TAF (or FTC/TDF + 3rd agent if currently or previously participated in Study GS-US-292-1826 [NCT02616783]) for the last 2 visits preceding the screening visit (or undetectable HIV-1 RNA level according to the local assay being used if the limit of detection is ≥ 50 copies/mL)
* Adequate renal function, an estimated glomerular filtration rate (eGFR) ≥ 30 mL/min according to the Cockcroft-Gault formula for creatinine clearance

Key Exclusion Criteria:

* An opportunistic illness indicative of stage 3 HIV diagnosed within the 30 days prior to screening
* Decompensated cirrhosis (eg, ascites, encephalopathy, or variceal bleeding)
* Current alcohol or substance use judged by the investigator to potentially interfere with participant study compliance

Note: Other protocol defined Inclusion/ Exclusion criteria may apply.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 86 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2020-05-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (25):
- Belgium (2):
  - CHU Saint-Pierre, Brussels
  - UZ Gent, Ghent
- France (9):
  - Hopital Saint-Andre, Bordeaux
  - Hopital Europeen Marseille, Marseille
  - C.H.U. de Nantes - Hotel Dieu, Nantes
  - CHU de Nice, Nice
  - Hopital Necker - Enfants Malades, Paris
  - Hopital Saint Louis, Paris
  - Hopital Saint Antoine, Paris
  - Interne et Maladies infectieuses, Pessac
  - CH de Tourcoing, Tourcoing
- Italy (4):
  - ASST Papa Giovanni XXIII, Bergamo
  - ASST - Fatebenefratelli Sacco, Milan
  - P.O. Spirito Santo - U.O. Malattie Infettive e Tropicali, Pescara
  - IRCCS Istituto Nazionale per le Malattie Infettive Lazzaro Spallanzani, Roma
- Spain (9):
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Costa Del Sol, Marbella
- Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified external researchers may request IPD for this study after study completion. For more information, please visit our website at https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy.
Supporting Information: Study Protocol, SAP
Time Frame: 18 months after study completion
Access Criteria: A secured external environment with username, password, and RSA code.
URL: https://www.gilead.com/science-and-medicine/research/clinical-trials-transparency-and-data-sharing-policy

REFERENCES:
- [Derived] Maggiolo F, Rizzardini G, Molina JM, Pulido F, De Wit S, Vandekerckhove L, Berenguer J, D'Antoni ML, Blair C, Chuck SK, Piontkowsky D, Martin H, Haubrich R, McNicholl IR, Gallant J. Bictegravir/emtricitabine/tenofovir alafenamide in older individuals with HIV: Results of a 96-week, phase 3b, open-label, switch trial in virologically suppressed people >/=65 years of age. HIV Med. 2023 Jan;24(1):27-36. doi: 10.1111/hiv.13319. Epub 2022 May 8. PMID 35527425
- [Derived] Maggiolo F, Rizzardini G, Molina JM, Pulido F, De Wit S, Vandekerckhove L, Berenguer J, D'Antoni ML, Blair C, Chuck SK, Piontkowsky D, Martin H, Haubrich R, McNicholl IR, Gallant J. Bictegravir/Emtricitabine/Tenofovir Alafenamide in Virologically Suppressed People with HIV Aged >/= 65 Years: Week 48 Results of a Phase 3b, Open-Label Trial. Infect Dis Ther. 2021 Jun;10(2):775-788. doi: 10.1007/s40121-021-00419-5. Epub 2021 Mar 9. PMID 33686573

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Europe. The first participant was screened on 01 March 2018. The last study visit occurred on 29 May 2020.
Pre-assignment Details: 90 participants were screened.
Groups:
- B/F/TAF: Bictegravir/emtricitabine/tenofovir alafenamide (B/F/TAF) (50/200/25 mg) fixed-dose combination (FDC) tablet once daily, without regard to food for at least 96 weeks.
Period: Overall Study
Arm/Group | B/F/TAF
Started | 86
Completed | 78
Not Completed | 8
Not completed — Adverse Event | 3
Not completed — Death | 2
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who were enrolled and received at least 1 dose of study drug.
Groups:
- B/F/TAF: B/F/TAF (50/200/25 mg) FDC tablet once daily, without regard to food for at least 96 weeks.
Arm/Group | B/F/TAF
Number analyzed (Participants) | 86
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (3.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 75
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not Permitted = Data not collected due to regional regulations or participant refused to provide information
  Participants
    Race: American Indian or Alaska Native | 0
    Race: Asian | 0
    Race: Black | 1
    Race: Native Hawaiian or Pacific Islander | 0
    Race: White | 82
    Race: Other | 0
    Race: Not Permitted | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not Permitted = Data not collected due to regional regulations or participant refused to provide information
  Participants
    Ethnicity: Hispanic or Latino | 12
    Ethnicity: Not Hispanic or Latino | 71
    Ethnicity: Not Permitted | 3
Region of Enrollment [Number; unit: participants]
  Belgium | 8
  France | 28
  Italy | 22
  Spain | 27
  United Kingdom | 1
Human Immunodeficiency Virus-1 Ribonucleic acid (HIV-1 RNA) Category [Count of Participants; unit: Participants]
  < 50 copies/mL | 84
  ≥ 50 copies/mL | 2
Cluster of Differentiation 4 (CD4) Cell Count [Mean (Standard Deviation); unit: cells/µL] | 694 (273.6)
CD4 Cell Count Category [Count of Participants; unit: Participants]
  < 50 cells/µL | 0
  ≥ 50 to < 200 cells/µL | 2
  ≥ 200 to < 350 cells/µL | 7
  ≥ 350 to < 500 cells/µL | 9
  ≥ 500 cells/µL | 68
CD4 Percentage [Mean (Standard Deviation); unit: percentage of lymphocytes] | 33.4 (9.24)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 24 as Defined by the Food and Drug Administration (FDA)-Defined Snapshot Algorithm
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 24 was analyzed using the snapshot algorithm, which defined a participant's virologic response status using only the viral load at the predefined timepoint within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 24
Population: The Full Analysis Set (FAS) included all participants who were enrolled and received at least 1 dose of study drug; and did not have major protocol violations.
Measure: Number; unit: percentage of participants
Arm/Group | B/F/TAF
Number analyzed (Participants) | 86
percentage of participants | 97.7

2. Secondary Outcome: Percentage of Participants Experiencing Adverse Events (AEs) Through Week 24
Description: An AE was any untoward medical occurrence in a clinical study participant administered a medicinal product, which did not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and/or unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. AEs may also included pre- or post-treatment complications that occurred as a result of protocol specified procedures, lack of efficacy, overdose, drug abuse/misuse reports, or occupational exposure. Preexisting events that increased in severity or changed in nature during or as a consequence of participation in the clinical study were also considered AEs.
Time Frame: First dose date up to Week 24
Population: The Safety Analysis Set included all participants who were enrolled and received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | B/F/TAF
Number analyzed (Participants) | 86
percentage of participants | 62.8

3. Secondary Outcome: Percentage of Participants Experiencing AEs Through Week 48
Description: as for outcome 2
Time Frame: First dose date Up to Week 48
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | B/F/TAF
Number analyzed (Participants) | 86
percentage of participants | 81.4

4. Secondary Outcome: Percentage of Participants Experiencing AEs Through Week 72
Description: as for outcome 2
Time Frame: First dose date Up to Week 72
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | B/F/TAF
Number analyzed (Participants) | 86
percentage of participants | 94.2

5. Secondary Outcome: Percentage of Participants Experiencing AEs Through Week 96
Description: as for outcome 2
Time Frame: First dose date Up to Week 96
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | B/F/TAF
Number analyzed (Participants) | 86
percentage of participants | 95.3

6. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 48 as Defined by the FDA-Defined Snapshot Algorithm
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 48 was analyzed using the snapshot algorithm, which defined a participant's virologic response status using only the viral load at the predefined timepoint within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 48
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | B/F/TAF
Number analyzed (Participants) | 86
percentage of participants | 90.7

7. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 72 as Defined by the FDA-Defined Snapshot Algorithm
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 72 was analyzed using the snapshot algorithm, which defined a participant's virologic response status using only the viral load at the predefined timepoint within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 72
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | B/F/TAF
Number analyzed (Participants) | 86
percentage of participants | 94.2

8. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 96 as Defined by the FDA-Defined Snapshot Algorithm
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 96 was analyzed using the snapshot algorithm, which defined a participant's virologic response status using only the viral load at the predefined timepoint within an allowed window of time, along with study drug discontinuation status.
Time Frame: Week 96
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | B/F/TAF
Number analyzed (Participants) | 86
percentage of participants | 74.4

9. Secondary Outcome: Change From Baseline in CD4 Cell Count at Week 24
Time Frame: Baseline, Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | B/F/TAF
Number analyzed (Participants) | 84
cells/µL | 20 (141.8)

10. Secondary Outcome: Change From Baseline in CD4 Cell Count at Week 48
Time Frame: Baseline, Week 48
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | B/F/TAF
Number analyzed (Participants) | 76
cells/µL | 8 (174.8)

11. Secondary Outcome: Change From Baseline in CD4 Cell Count at Week 72
Time Frame: Baseline, Week 72
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | B/F/TAF
Number analyzed (Participants) | 78
cells/µL | 36 (145.7)

12. Secondary Outcome: Change From Baseline in CD4 Cell Count at Week 96
Time Frame: Baseline, Week 96
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: cells/µL
Arm/Group | B/F/TAF
Number analyzed (Participants) | 59
cells/µL | 22 (150.9)

13. Secondary Outcome: Change From Baseline in CD4 Percentage at Week 24
Time Frame: Baseline, Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of lymphocytes
Arm/Group | B/F/TAF
Number analyzed (Participants) | 84
percentage of lymphocytes | 0.1 (3.52)

14. Secondary Outcome: Change From Baseline in CD4 Percentage at Week 48
Time Frame: Baseline, Week 48
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of lymphocytes
Arm/Group | B/F/TAF
Number analyzed (Participants) | 76
percentage of lymphocytes | 0.1 (3.89)

15. Secondary Outcome: Change From Baseline in CD4 Percentage at Week 72
Time Frame: Baseline, Week 72
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of lymphocytes
Arm/Group | B/F/TAF
Number analyzed (Participants) | 78
percentage of lymphocytes | -0.1 (4.29)

16. Secondary Outcome: Change From Baseline in CD4 Percentage at Week 96
Time Frame: Baseline, Week 96
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of lymphocytes
Arm/Group | B/F/TAF
Number analyzed (Participants) | 59
percentage of lymphocytes | -0.1 (4.34)

17. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 24, as Analyzed by Missing = Failure Approach
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 24 was analyzed using missing = failure approach. In this approach, all missing data were treated as HIV-1 RNA ≥ 50 copies/mL.
Time Frame: Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | B/F/TAF
Number analyzed (Participants) | 86
percentage of participants | 97.7

18. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 48, as Analyzed by Missing = Failure Approach
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 48 was analyzed using missing = failure approach. In this approach, all missing data were treated as HIV-1 RNA ≥ 50 copies/mL.
Time Frame: Week 48
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | B/F/TAF
Number analyzed (Participants) | 86
percentage of participants | 90.7

19. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 72, as Analyzed by Missing = Failure Approach
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 72 was analyzed using missing = failure approach. In this approach, all missing data were treated as HIV-1 RNA ≥ 50 copies/mL.
Time Frame: Week 72
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | B/F/TAF
Number analyzed (Participants) | 86
percentage of participants | 94.2

20. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 96, as Analyzed by Missing = Failure Approach
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 96 was analyzed using missing = failure approach. In this approach, all missing data were treated as HIV-1 RNA ≥ 50 copies/mL.
Time Frame: Week 96
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | B/F/TAF
Number analyzed (Participants) | 86
percentage of participants | 79.1

21. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 24, as Analyzed by Missing = Excluded Approach
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 24 was analyzed using missing = excluded approach. In this approach, all missing data were excluded in the computation of the percentages (ie, missing data points were excluded from both the numerator and denominator in the computation).
Time Frame: Week 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | B/F/TAF
Number analyzed (Participants) | 84
percentage of participants | 100.0

22. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 48, as Analyzed by Missing = Excluded Approach
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 48 was analyzed using missing = excluded approach. In this approach, all missing data were excluded in the computation of the percentages (ie, missing data points were excluded from both the numerator and denominator in the computation).
Time Frame: Week 48
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | B/F/TAF
Number analyzed (Participants) | 78
percentage of participants | 100.0

23. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 72, as Analyzed by Missing = Excluded Approach
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 72 was analyzed using missing = excluded approach. In this approach, all missing data were excluded in the computation of the percentages (ie, missing data points were excluded from both the numerator and denominator in the computation).
Time Frame: Week 72
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | B/F/TAF
Number analyzed (Participants) | 81
percentage of participants | 100.0

24. Secondary Outcome: Percentage of Participants With HIV-1 RNA < 50 Copies/mL at Week 96, as Analyzed by Missing = Excluded Approach
Description: The percentage of participants with HIV-1 RNA < 50 copies/mL at Week 96 was analyzed using missing = excluded approach. In this approach, all missing data were excluded in the computation of the percentages (ie, missing data points were excluded from both the numerator and denominator in the computation).
Time Frame: Week 96
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | B/F/TAF
Number analyzed (Participants) | 68
percentage of participants | 100.0

ADVERSE EVENTS:
Time Frame: Adverse Events: First dose of study drug up to last dose plus 30 days (up to Week 102.9); All-Cause Mortality: First dose date up to Week 102.9
Description: The Safety Analysis Set included all participants who were enrolled and received at least 1 dose of study drug.
Arm/Group | B/F/TAF
All-Cause Mortality (participants affected / at risk) | 2/86
Serious Adverse Events (participants affected / at risk) | 9/86
Other Adverse Events (participants affected / at risk) | 34/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | B/F/TAF (N=86)
Atrial fibrillation (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 1
Anal abscess (Infections and infestations) | 1
Covid-19 pneumonia (Infections and infestations) | 1
Endocarditis (Infections and infestations) | 1
Intentional overdose (Injury, poisoning and procedural complications) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Ischaemic stroke (Nervous system disorders) | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 1
Completed suicide (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Suicide attempt (Psychiatric disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | B/F/TAF (N=86)
Diarrhoea (Gastrointestinal disorders) | 6
Bronchitis (Infections and infestations) | 10
Nasopharyngitis (Infections and infestations) | 7
Urinary tract infection (Infections and infestations) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 8
Sciatica (Nervous system disorders) | 5
Hypertension (Vascular disorders) | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2018-12-18): https://cdn.clinicaltrials.gov/large-docs/35/NCT03405935/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-19): https://cdn.clinicaltrials.gov/large-docs/35/NCT03405935/SAP_002.pdf